CLINICAL TRIAL: NCT04852874
Title: Is Quadratus Lumborum Block an Efficient and Safe Anesthetic Method for Percutaneous Nephrolithotomy? A Feasibility Study
Brief Title: Quadratus Lumborum Block as an Anesthetic Method for Percutaneous Nephrolithotomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abul-fotouh Ahmed, Professor of Urology and Andrology, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Uro_Azhar_8_021
Record Dates: First submitted 2021-04-09; First posted 2021-04-21 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Quadratus Lumborum Block; Percutaneous Nephrolithotomy; Local Anesthesia

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, open-label, interventional study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ultrasound-guided Quadratus Lumborum Block (Experimental)
  Interventions: Procedure: Ultrasound-guided Quadratus Lumborum Block

INTERVENTIONS:
Procedure: Ultrasound-guided Quadratus Lumborum Block — Low dose spinal anesthesia will be done at L3-4 lumbar vertebrae with bupivacaine 2.5 mg (0.5 ml Marcaine 0.5%) and fentanyl 25 µgm (0.5 ml) of fentanyl amp (100 µgm/ 2ml) to be added to 1.5 - 2 ml of free water to form total volume of 2.5- 3ml according to the patient height aiming level of T6 sensory level.
  Quadratus lumorum block:
  After 4 to 5 minutes, ultrasound guided quadratus lumborum block (QL 1,2,3) will be done unilaterally, using low-frequency convex probe, taking into consideration the total volume of injectate not exceeding 0.4 ml /kg of (bupivacaine 0.5%) to avoid local anesthesia systemic toxicity. This is equal to 0.8 ml/kg of (bupivacaine 0.25%).
  After confirming the correct position of the needle, 0.2-3 ml/kg of 0.25% bupivacaine plus 1.5 mg dexamethasone and magnesium sulphate of 100 mg will be injected in each site of the QL 1,2,3 using the lean body weight. The lean body weight will be calculated by omni lean body mass online calculator.

SUMMARY:
The study aims to investigate the efficacy and safety of QLB, as an anaesthetic method, for patients undergoing PCNL. Adult patients who agree to participate in the study will be included. Uncooperable patients, pregnant woman, active urinary tract infection, uncorrectable coagulation disorder, and those with known allergy to study medication will be excluded. Low dose spinal anaesthesia and Ultrasound-guided QLB will be performed. The success of the procedure, procedure-related complications, Intra- and post-operative hemodynamics, pain score, overall surgeon and patient satisfaction will be evaluated and reported.

DETAILED DESCRIPTION:
Percutaneous nephrolithotomy (PCNL) is used more frequently than open surgery in the treatment of kidney stones as it is performed through a smaller surgical incision. Postoperative complex pain resulting from the renal capsule dilation and nephrostomy-tube-related stress is reported to prolong the recovery time, reduce patient comfort, and increase complication rates. Opioids, which are used for controlling Intra and postoperative pain, have significant side effects. Multi-modal analgesia regimen and regional anaesthesia methods have been reported to decrease the side effects, in addition to providing effective postoperative pain control.

The use of an intraoperative local anaesthetic or peripheral blocks as an analgesic has been reported for pain control in PCNL but only as analgesia not anaesthesia except loco-regional like spinal and epidural anaesthesia with limitation of time or cardiopulmonary side effects that usually in favour of general anaesthesia that is usually considered the most convenient and prudent way for providing anaesthesia for this operation in spite of its drawbacks.

The quadratus lumborum muscle block (QLB) was first described by Blanco in 2007 as a local anaesthetic injection into the anterolateral junction of the quadratus lumborum muscle (QLB type 1). QLB does not only stop somatic pain but also it inhibits visceral pain due to the spread of the local anaesthetic to the paravertebral space.

Some modifications of this technique were subsequently introduced: injection into the posterior segment of the quadratus lumborum muscle (QLB type2), injection between the quadratus lumborum muscle and the fascia of the psoas muscle using the trans muscular approach (QLB type 3), and injection into the quadratus lumborum muscle (QLB type 4) itself. It is evident that this block is effective in providing analgesia from T7 to L1 dermatomes, it is not only providing analgesia from the anterior abdominal wall but also it can reduce visceral pain.

Although the efficacy of QLB in abdominal surgery has been demonstrated in the literature, its use as an anaesthesia technique not ever reported.

In this study, the investigators introduce a new protocol in providing anaesthesia mainly by fascial peripheral block. It is considered new as it is the first time to our knowledge to use a fascial block as a main component of anaesthesia for PCNL and the investigators think that it may be used as a solo anaesthesia. This will lead to decreasing patient stay in the hospital, decreasing time for patient ambulation and regaining vitality and hemostasis that will all be in line with early rehabilitation after surgery (ERAS) protocol that is the aim of all health care services in modern medicine. Also, it will be the base for further research in more risky patient groups that may decrease the detrimental effect of general anaesthesia in these patient group which already have associated comorbidities and for more operation especially if unilateral.

In this study, the investigators will evaluate the efficacy and safety of ultrasound-guided QLB as an anaesthetic method in patients undergoing PCNL.

Adult patients who will undergo elective unilateral PCNL will be included. Low dose spinal anaesthesia will be done at L3-4 lumbar vertebrae. Then, ultrasound-guided QLB (QL 1,2,3) will be performed on the ipsilateral surgical side, using a low-frequency convex transducer. The total volume of injectate will not exceed 0.4 ml /kg of (bupivacaine 0.5%).

The success of the procedure, procedure-related complications, Intra- and post-operative hemodynamics, pain score, overall surgeon and patient satisfaction will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients who will undergo an elective unilateral PCNL and agree to participate in the study will be included

Exclusion Criteria:

* Uncooperable patients
* Pregnant women
* Untreated urinary tract infection
* Uncorrected coagulation disorder
* Known allergy to study medications
* Local infection at the site of injection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2021-04-03 (Actual); Primary Completion 2023-04-01 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
Success of the QLB | At the end of PCNL procedure.
  Accomplishing of the PCNL procedure with no need of alteration to general anesthesia with neutral or more better levels of surgeon and patient satisfaction using a five-point scale of customer Satisfaction survey score of 5 points

SECONDARY OUTCOMES:
Blood pressure | Intra-operative
Pulse | Intra-operative
spo2 | Intra-operative
Visual analogue scale | Intra-operative, and post-operative at 0,1,2, 4, 8, 12,16,20,24 hours
  0-to-10 scale, where 0 (no pain) and 10 (worst imaginable pain).
Time for the 1st analgesic requirement. | Intra- and post-operative up to 24 hours
  The time from performance the block until the patient asked analgesia with visual analogue visual analogue pain scale ≥ 4
QLB-related complications | Intra- and post-operative up to 24 hours
  e.g of hypotension related to block, defined as decreases in mean arterial blood pressure more than 20% of the basal BP
Patient's satisfaction | Intra- and post-operative, up to 24 hours
  A five-point scale will be used to asses satisfaction, where 1 is unsatisfied and 5 fully satisfied.
Surgeon's satisfaction | Intra- and post-operative up to 24 hours
  A five-point scale will be used to asses satisfaction, where 1 is unsatisfied and 5 fully satisfied.
PCNL complications | up to 3 months
Need for ancillary procedure | up to 3 months
Stone free rate | up to 3 months post-operative
  stone-free status is defined as no stones or residual fragment less than 4 mm on NCCT

CONTACTS AND LOCATIONS:
Locations (1):
- Urology Department, Al-Azhar University Hospital, Cairo, Egypt